CLINICAL TRIAL: NCT05813145
Title: Fenofibrate Role Against Chemotherapy Induced Peripheral Neurotoxicity in Breast Cancer Patients
Brief Title: Fenofibrate Role in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fenofibrate in Breast Cancer
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: Group 1 ( Arm A) (n=25: will receive four cycle of AC followed by paclitaxel 80 mg/m2 weekly for 12 week.
  Group 2 ( Arm B) (n=25): will receive the same regimen as group1 in addition to 160mg (17 ,18 ) fenofibrate once daily for 3 month.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): n=25: will receive Placebo plus four cycle of AC followed by paclitaxel 80 mg/m2 weekly for 12 week.
  Interventions: Drug: Placebo
- fenofibrate group (Active Comparator): n=25: will receive fenofibrate 160mg once daily for 3 month plus four cycle of AC followed by paclitaxel 80 mg/m2 weekly for 12 week.
  .
  Interventions: Drug: Fenofibrate 160mg

INTERVENTIONS:
Drug: Placebo — 25 patients will receive four cycle of AC followed by paclitaxel 80 mg/m2 weekly for 12 week
  Other Names: Placebo tablet
  Arms: Placebo Group
Drug: Fenofibrate 160mg — 25 patients will receive four cycle of AC followed by paclitaxel 80 mg/m2 weekly for 12 week in addition to 160mg fenofibrate once daily for 3 month.
  Other Names: Lipanthyl 16omg
  Arms: fenofibrate group

SUMMARY:
The aim of the study is to assess the efficacy of fenofibrate in either reversing and/or preventing the development of PIPN in breast cancer patients treated with paclitaxel-based regimen. The primary outcome :clinical improvement of neuropathic pain and grade by 1-CT-CTCAE -VERSION-4 & FACT/GOG-NT-12 questionnaire and its effect on quality of life (QOL).

The secondary outcome : the efficacy of fenofibrate in either reversing and/or preventing the development of PIPN via alteration of either Nerve growth factor (NGF) or/ and/( NFL).

DETAILED DESCRIPTION:
Ethical committee approval will be obtained from ethics committee of Faculty of Pharmacy, Damanhur University.

2. All participants should agree to take part in this clinical study and will provide informed consent.

3. fifty female patients with diagnosed breast cancer, who are candidates for will be recruited from Damanhur oncology center.

4. All enrolled patients will be randomly assigned into two arms: Group 1 ( Arm A) (n=25: will receive four cycle of AC followed by paclitaxel 80 mg/m2 weekly for 12 week.

Group 2 ( Arm B) (n=25): will receive the same regimen as group1 in addition to 160mg (17 ,18 ) fenofibrate once daily for 3 month.

5. All patients will be submitted to:

* Full patient history and clinical examination.
* Routine follow up before and after each chemotherapy cycle (complete blood picture, liver function tests, renal function tests).
* Serum samples will be collected from patients at the time of admission for measuring the neuropathy biomarkers Nerve growth factor (NGF) and (NFL) to lipid profile .
* Clinical assessment of neuropathic pain using FACT/GOG NtX 12 questionnaire and NCT-CTCAE -VERSION-4 .

  6. All patients will be followed up during paclitaxel treatment period (12 weeks). At the end of paclitaxel treatment, Serum samples will be collected from patients for measuring the biomarkers .

  7. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.

  8. Results, conclusion, discussion, and recommendations will be given.

ELIGIBILITY:
Inclusion criteria:

1. included a diagnosis breast cancer with age > 18 years.
2. Naïve to chemotherapy

Exclusion Criteria:

1. Concurrent administration (statins , cyclosporine) .
2. Advanced liver disease (defined as liver enzyme elevation >3-fold upper limit of normality, or cirrhosis); chronic kidney disease (CKD, defined as an eGFR <60 ml min-1 1.73 m-2); acute or chronic pancreatitis and diabetes.
3. Patients with a history of allergy to fenofibrate.
4. Concomitant use of opioids, anticonvulsants, tricyclic antidepressants, other neuropathic pain medication.
5. Pregnancy or breast feeding.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Nerve growth factor (NGF) Concentration | 3 month
  Concentration of Nerve growth factor (NGF)
Neurofilament light chain (NfL) protein Concentration | 3 month
  Concentration of Neurofilament light chain (NfL) protein

SECONDARY OUTCOMES:
Incidence of neuropathic pain | 6 months
  neuropathic pain using score from FACT/GOG NtX 12 questionnaire .

CONTACTS AND LOCATIONS:
Overall Officials: Noha El bassiouny, Lecturer, Study Director — Damanhour University
Locations (1):
- Damanhour Oncology Center, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Othman A, Benghozi R, Alecu I, Wei Y, Niesor E, von Eckardstein A, Hornemann T. Fenofibrate lowers atypical sphingolipids in plasma of dyslipidemic patients: A novel approach for treating diabetic neuropathy? J Clin Lipidol. 2015 Jul-Aug;9(4):568-75. doi: 10.1016/j.jacl.2015.03.011. Epub 2015 Apr 4. PMID 26228675
- [Background] Caillaud M, Patel NH, White A, Wood M, Contreras KM, Toma W, Alkhlaif Y, Roberts JL, Tran TH, Jackson AB, Poklis J, Gewirtz DA, Damaj MI. Targeting Peroxisome Proliferator-Activated Receptor-alpha (PPAR- alpha) to reduce paclitaxel-induced peripheral neuropathy. Brain Behav Immun. 2021 Mar;93:172-185. doi: 10.1016/j.bbi.2021.01.004. Epub 2021 Jan 9. PMID 33434562